CLINICAL TRIAL: NCT05641441
Title: Radiosurgery Induced Ototoxicity in Patients Treated for a Vestibular Schwannoma
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Pascal Senn, Chairman of the Service of Otorhinolaryngology-Head and Neck Surgery, Department of clinical neurosciences, Geneva University Hospitals, University Hospital, Geneva
Other Study IDs: 2022-01257
Record Dates: First submitted 2022-11-16; First posted 2022-12-07 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Vestibular Schwannoma; Ototoxicity
Keywords: Radiosurgery; Ototoxicity; Vestibular Schwannoma; Hearing loss; Quality of Life
MeSH Terms: conditions — Neuroma, Acoustic; Ototoxicity; Hearing Loss | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stereotactic radiosurgery group: Patients with unilateral Vestibular Schwannoma treated with stereotactic radiosurgery, as proposed by the institution's skull base tumor board independently of the study.
  Interventions: Radiation: Stereotactic radiosurgery
- Wait and scan group: Patients with unilateral Vestibular Schwannoma followed with an MRI-based observation strategy, as proposed by the institution's skull base tumor board independently of the study.

INTERVENTIONS:
Radiation: Stereotactic radiosurgery — Stereotactic radiosurgery
  Groups: Stereotactic radiosurgery group

SUMMARY:
The investigators aim to study the impact of stereotactic radiosurgery, for the treatment of vestibular Schwannoma, on the cochlear, vestibular, gustatory, and facial nerve functions and compare it with a conservatively treated group. The predictive value of radiological tumor characteristics on hearing preservation and vestibular function will be also evaluated.

Additionally, the investigators will invite patients with vestibular Schwannoma to fill out questionnaires to assess their quality of life.

DETAILED DESCRIPTION:
The study will have a retrospective part and a prospective part. The retrospective study will be based on a series of consecutive patients with vestibular Schwannoma (VS) treated either with stereotactic radiosurgery (SRS) or followed up radiologically between 2014 and 2021 in our institution. The following data will be retrieved from the hospital archiving system and will be subsequently analyzed: demographics, patient characteristics, details regarding SRS planning, clinical baseline and follow-up data, hearing, vestibular and taste function assessment initially and during follow-up, presence of additional symptoms (tinnitus, hemifacial spasm, trigeminal neuralgia), radiosurgery parameters and MRI characteristics of tumors. The following parameters will be retrospectively measured on MRI images by an experienced radiologist in each VS: tumor volume, ratio of brain stem compression, tumor shape and distance to the fundus of the internal auditory canal, length of the tumor in the internal auditory canal, and signal intensity in the cochlea and vestibule. The MRI textural features extracted from whole tumor segmentation of VSs will be calculated and analyzed with MatLab®. They include shape features, first order and second order textural features.

The prospective study part aims to obtain more precise and predefined follow-up data from patients treated either with SRS or followed up conservatively from now on. Our institution's multidisciplinary skull base tumor board will be responsible for treatment decisions independently of the study. It will be a single-center observational cohort study investigating the respective impact of tumor morphology and SRS on the inner ear, the facial nerve function, and the quality of life of these patients. As data collection will be done prospectively, MRI acquisition parameters will be standardized, as well as quantification of hearing, vestibular, facial nerve function, and quality of life. Additionally, the investigators will analyze the characteristics of the tumors and several parameters of the irradiation protocol to develop predictive models for ototoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* Patients with unilateral VS treated either with SRS or MRI-based observation strategy, as proposed by the institution's skull base tumor board independently of the study
* Patients willing to take part in the study and give their informed consent

Exclusion Criteria:

* Previous surgical or radiation therapy for VS (including SRS)
* Patients diagnosed with neurofibromatosis type II
* Preexisting profound hearing loss, with a pure tone average (PTA) >90 and word recognition score (WRS) <10%, upon initial assessment
* Previous middle ear surgery of the affected ear
* Concurrent treatment with other experimental drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at the Geneva University Hospitals (tertiary care facility) in Switzerland. For the retrospective part of our research project, the investigators aim to analyze non-genetic health-related personal data in a coded form from approximately 150 patients treated between 2014 and 2021.
  Regarding the prospective study part, patient recruitment will be done through the multidisciplinary skull base tumor board, where cases are discussed in detail, treatment decisions are made consensually based on the contribution of different specialists and in agreement with the current international recommendations. Patients eligible for study inclusion will be contacted to obtain informed consent. The investigators aim to include 108 participants.
Sampling Method: Probability Sample
Enrollment: 258 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2030-11-15 (Estimated); Study Completion 2030-11-15 (Estimated)

PRIMARY OUTCOMES:
Change of Pure Tone Average from baseline | 1-year
  Hearing status as measured by audiometric tonal testing and calculated from the average of 500 Hz, 1000 Hz, 2000 Hz and 3000 Hz.
Change of Word recognition score from baseline | 1-year
  Hearing status as measured by audiometric vocal testing and calculated as the percentage of correctly identified monosyllabic words presented at the speech recognition threshold + 40 decibel hearing level

SECONDARY OUTCOMES:
Change of Pure Tone Average from baseline | 3 and 5-year
  Hearing status as measured by audiometric tonal testing and calculated from the average of 500 Hz, 1000 Hz, 2000 Hz and 3000 Hz.
Change of High-frequency Pure Tone Average from baseline | 1, 3 and 5-year
  Hearing status as measured by audiometric tonal testing and calculated from the average of 3000 Hz, 4000 Hz and 6000 Hz.
Change of Word recognition score from baseline | 3 and 5-year
  Hearing status as measured by audiometric vocal testing and calculated as the percentage of correctly identified monosyllabic words presented at the speech recognition threshold + 40 decibel hearing level
Change of video-oculography from the baseline | 1, 3 and 5-year
  Video-oculography assessment to detect a pathologic nystagmus or a pathologic smooth pursuit
Change of caloric ipsilateral testing (degree of asymmetry) from baseline | 1, 3 and 5-year
  Caloric testing to assess the vestibulo-ocular reflex in the low-frequency range.
Change of the cervical Vestibular Evoked Myogenic Potential (cVEMP) from baseline | 1, 3 and 5-year
  Assessment of a present or absent reflex which reflects the function of saccule
Change of the ocular Vestibular Evoked Myogenic Potential (oVEMP) from baseline | 1, 3 and 5-year
  Assessment of a present or absent reflex which reflects the function of utricle
Change of the Video Head Impulse Test (VHIT) from baseline | 1, 3 and 5-year
  Assessment of the VHIT to detect dysfunction of the vestibulo-ocular reflex in the high-frequency range.
Change of facial nerve function from baseline | 1, 3 and 5-year
  House-Brackmann scale score ranges from 1 (best) to 6 (worst)
Change of taste function from baseline | 6 and 12-month
  "Taste strips" test score ranges from 0 (worst) to 16 (best) on each side of the tongue
Change of 36-Item Short Form Health Survey (SF-36) score from baseline | 1, 3 and 5-year
  SF-36 score ranges from 0 (worst) to 100 (best)
Change of Penn Acoustic Neuroma Quality-of-Life (PANQOL) scale score from baseline | 1, 3 and 5-year
  Penn Acoustic Neuroma Quality-of-Life (PANQOL) scale score ranges from 0 (worst) to 100 (best)
Change of Tinnitus Handicap Inventory (THI) score from baseline | 1, 3 and 5-year
  Tinnitus Handicap Inventory (THI) score ranges from 0 (best) to 100 (worst)

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ORL et Chirurge cervico-faciale, Hopitaux Universitaires de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://recherche.hug.ch/etudes/etude-clinique-sur-le-schwannome-vestibulaire